CLINICAL TRIAL: NCT05347394
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single- and Multiple-dose Escalation Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of Oral VX-708 in Healthy Subjects
Brief Title: A Phase 1 Dose Escalation Study of Oral VX-708 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX21-708-002; 2021-005559-35 (EudraCT Number)
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: VX-708 (Experimental): Participants will be randomized to receive a single dose of different dose levels of VX-708.
  Interventions: Drug: VX-708
- Part A: Placebo (Placebo Comparator): Participants will receive placebo matched to VX-708.
  Interventions: Drug: Placebo
- Part B: VX-708 (Experimental): Participants will be randomized to receive multiple doses of different dose levels of VX-708. The dose levels will be determined based on the data from Part A.
  Interventions: Drug: VX-708
- Part B: Placebo (Placebo Comparator): Participants will receive placebo matched to VX-708.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-708 — Solution or suspension for oral administration.
  Arms: Part A: VX-708; Part B: VX-708
Drug: Placebo — Placebo matched to VX-708 for oral administration.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple ascending doses of VX-708 in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female of non-childbearing potential are eligible
* Body mass index (BMI) of 18.0 to 32.0 kilograms per meter square (kg/m^2)
* A total body weight greater than (>) 50 kg

Key Exclusion Criteria:

* History of febrile illness or other acute illness within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption, distribution, metabolism, or excretion
* History of cardiac dysrhythmias

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 25
Part B: Safety and Tolerability as Assessed by Number of Participants With Clinically Meaningful Findings in Columbia Suicide Severity Rating Scale (C-SSRS) Responses | From Day 1 up to Day 25

SECONDARY OUTCOMES:
Parts A and B: Area Under the Plasma Concentration Versus Time Curve During a Dosing Interval (AUCtau) of VX-708 | From Day 1 up to Day 25
Part B: Pain Tolerance Threshold (PTT) for the Cold Pressor Test | From Day 1 up to Day 11

CONTACTS AND LOCATIONS:
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing